CLINICAL TRIAL: NCT02994784
Title: A Phase II Single-Center, Open-Label, Safety and Efficacy Study of Propylene Glycol-Free Melphalan Hydrochloride (Evomela) in AL Amyloidosis Patients Undergoing Autologous Stem Cell Transplantation
Brief Title: Propylene Glycol-Free Melphalan Hydrochloride (Evomela) in AL Amyloidosis Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual during COVID pandemic, alternative treatments available. Study halted early.
Sponsor: Boston Medical Center (Other)
Collaborators: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-35835
Record Dates: First submitted 2016-11-18; First posted 2016-12-16 (Estimated); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Amyloidosis; Systemic
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evomela (Experimental): Propylene Glycol-Free Melphalan Hydrochloride (Evomela) administered intravenously at 70-100 mg/m2/day on Days -3 and -2 prior to autologous stem cell transplantation
  Interventions: Drug: Propylene Glycol-Free Melphalan Hydrochloride

INTERVENTIONS:
Drug: Propylene Glycol-Free Melphalan Hydrochloride — Intravenous Propylene Glycol-Free Melphalan Hydrochloride
  Other Names: Evomela

SUMMARY:
This is a single arm, open label study designed to evaluate the safety and efficacy of propylene glycol-free melphalan hydrochloride in patients with AL amyloidosis. Treatment will be comprised of propylene glycol-free melphalan hydrochloride administered intravenously at a dose of 70-100 mg/m2/day on Days -3 and -2 as conditioning prior to autologous stem cell transplantation.

DETAILED DESCRIPTION:
After giving written informed consent, subjects will be evaluated for eligibility for enrollment in the study. Baseline evaluations will be performed as outlined in Section 7. Subjects who satisfy all inclusion and exclusion criteria will begin the study drug. Subjects will be monitored from the time of the medication administration until discharge from the transplant program for safety. Organ function and hematologic status will also be measured at 6 and 12 month follow-up visits.

Standard response criteria for AL amyloidosis hematologic and organ response will be used. Overall response rate will be measured and participants will be categorized into complete response, very good partial response, partial response and progressive disease. Progression free survival, organ response, and safety and tolerability of propylene glycol-free melphalan hydrochloride will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Eastern Cooperative Oncology Group Performance Status 0-2
* Histologic diagnosis of primary systemic (AL) amyloidosis based on:

  * Deposition of amyloid material by Congo red stain showing characteristic apple green birefringence AND
  * Evidence of a clonal plasma cell dyscrasia with monoclonal protein in the serum or urine by immunofixation electrophoresis AND/OR abnormal serum free light chain assay AND/OR clonal plasma cells in the bone marrow exam demonstrated by immunohistochemistry, flow cytometry, or in situ hybridization AND
  * Evidence of organ involvement
* Eligible for treatment with high dose melphalan and stem cell transplantation per institutional guidelines
* Ability to understand and willingness to sign informed consent
* Pulmonary Function Test demonstrating a diffusion capacity of lung for carbon monoxide ≥ 50%
* Left ventricular ejection fraction ≥40%
* Systolic blood pressure >90 mm Hg (supine position)
* Eastern Cooperative Oncology Group Performance status of 2 or better (unless patient is diagnosed with AL amyloidosis involving the gastrointestinal and peripheral/autonomic nervous systems, then performance status of 3 is acceptable)

Exclusion Criteria:

* Previous high-dose melphalan and stem cell transplant
* Previous total cumulative dose of oral melphalan > 300 mg
* Cytotoxic chemotherapy within the previous 28 days
* New York Heart Association ≥3
* Decompensated or uncontrolled heart failure
* Oxygen dependence
* epidermal growth factor receptor < 30 ml/min
* Active infection (i.e HIV, Hepatitis B or C)
* Pregnancy or breastfeeding
* Exposure to another investigational drug within 3-4 weeks prior to start of study treatment
* Ongoing alcohol or drug addiction
* Unable or unwilling to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Sloan, MD, Principal Investigator — Attending Physician
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data.

REFERENCES:
- [Background] Palladini G, Dispenzieri A, Gertz MA, Kumar S, Wechalekar A, Hawkins PN, Schonland S, Hegenbart U, Comenzo R, Kastritis E, Dimopoulos MA, Jaccard A, Klersy C, Merlini G. New criteria for response to treatment in immunoglobulin light chain amyloidosis based on free light chain measurement and cardiac biomarkers: impact on survival outcomes. J Clin Oncol. 2012 Dec 20;30(36):4541-9. doi: 10.1200/JCO.2011.37.7614. Epub 2012 Oct 22. PMID 23091105
- [Derived] Sarosiek S, Lee MH, Doros G, Edwards CV, Quillen K, Brauneis D, Shelton AC, Sanchorawala V, Sloan JM. Safety and Efficacy of Propylene Glycol-Free Melphalan in Patients with AL Amyloidosis Undergoing Autologous Stem Cell Transplantation: Results of a Phase II Study. Transplant Cell Ther. 2023 Nov;29(11):695.e1-695.e7. doi: 10.1016/j.jtct.2023.08.018. Epub 2023 Aug 20. PMID 37607644

RESULTS

PARTICIPANT FLOW:
Period: Enrolled
Arm/Group | Evomela
Started | 27
Completed | 27
Not Completed | 0
Period: 6 Months Follow-up
Arm/Group | Evomela
Started | 27
Completed | 24
Not Completed | 3
Not completed — Lost to Follow-up | 3
Period: 12 Month Follow-up
Arm/Group | Evomela
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Evomela
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 60 [44 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 20
  Black | 6
  Asian | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Renal Dysfunction
Description: To determine the safety profile of propylene glycol-free melphalan hydrochloride in the conditioning regimen prior to autologous stem cell transplantation in AL amyloidosis patients, including adverse events related to renal dysfunction (was acute renal failure is defined as either a >/=1 mg/dL increase in serum creatinine or a doubling of serum creatinine to >/=1.5 mg/dL for at least 2 days.).
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Evomela
Number analyzed (Participants) | 27
Participants | 2

2. Primary Outcome: Number of Participants With Cardiac Dysfunction (New Arrhythmia)
Description: To determine the safety profile of propylene glycol-free melphalan hydrochloride in the conditioning regimen prior to autologous stem cell transplantation in AL amyloidosis patients, including adverse events related to cardiac dysfunction (new arrhythmia).
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Evomela
Number analyzed (Participants) | 27
Participants | 5

3. Secondary Outcome: Neutrophil Engraftment
Description: time to neutrophil engraftment
Time Frame: 3 weeks
Measure: Median (Full Range); unit: days
Arm/Group | Evomela
Number analyzed (Participants) | 27
days | 10 [8 to 14]

4. Secondary Outcome: Platelet Engraftment
Description: Assess time to platelet engraftment
Time Frame: 100 days
Measure: Median (Full Range); unit: days
Arm/Group | Evomela
Number analyzed (Participants) | 27
days | 17 [14 to 27]

5. Secondary Outcome: Treatment Related Mortality
Description: Number of patients who expire within 100 days of transplant
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Evomela
Number analyzed (Participants) | 27
Participants | 0

6. Secondary Outcome: Hematologic Overall Response Rate
Description: Number of patients with response based on Gertz, Palladini criteria (below) Complete response (CR): Normal serum free light chain ratio,Negative serum and urine immunofixation electrophoresis Very good partial response (VGPR): Difference in serum free light chains less than 40 mg/L Partial Response (PR): >50% Reduction in the difference in serum free light chains Stable Disease (SD): Meets neither criteria for CR, VGPR, PR or PD
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Evomela
Number analyzed (Participants) | 27
Participants | 22

7. Secondary Outcome: Organ Response
Description: Number of patients with organ response based on Gertz criteria (below)
  * Kidney: 50% reduction in 24-hour urine protein excretion in the absence of progressive renal insufficiency (defined as a 25% increase in serum creatinine, as long as that is > to an absolute increase of 0.5 mg/dL). In the case of nephrotic syndrome: a decrease in proteinuria to < 1g/24h and an improvement in one of 2 extrarenal features - normalization of serum albumin or resolution of edema and/or discontinuation of diuretics in response to improvement in edema.
  * Heart: ≥ 2 mm reduction in the interventricular septal (IVS) thickness by echocardiogram, improvement of ejection fraction by ≥ 20% (echocardiogram must be performed at the same institution), or decrease in 2 NYHA classes without increase in diuretic need.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Evomela
Number analyzed (Participants) | 24
Participants | 13

8. Secondary Outcome: Participants With Peri-transplant Hospitalizations
Description: Number of participants with peri-transplant hospitalizations
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Evomela
Number analyzed (Participants) | 27
Participants | 23

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Evomela
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 20/27
Other Adverse Events (participants affected / at risk) | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evomela (N=27)
Cardiac arrhythmias (Cardiac disorders) | 4 (4) — New cardiac arrhythmias
Renal dysfunction (Renal and urinary disorders) | 2 (2)
Autonomic dysfunction (Nervous system disorders) | 14 (14)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evomela (N=27)
Diarrhea (Gastrointestinal disorders) | 25 (25)
Nausea (Gastrointestinal disorders) | 20 (20)
Fatigue (General disorders) | 22 (22)

LIMITATIONS AND CAVEATS:
Study was halted early resulting in relatively small numbers of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT02994784/Prot_SAP_000.pdf